CLINICAL TRIAL: NCT03901989
Title: Treatment of Osteoporosis by Panaceo: Randomized, Double-blind, Controlled, Study Assessed Effect on Bone Mineral Density and Bone Turnover of Panaceo Compared to Placebo in Osteoporotic Patients
Brief Title: Treatment of Osteoporosis - TOP1 Clinical Study
Acronym: TOP1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinic K-center (Other)
Collaborators: University of Rijeka (Other)
Responsible Party: Principal Investigator, DALIBOR KRPAN, Prof.dr.sc. Dalibor Krpan, prim.dr.med., Polyclinic K-center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TOP 001-2013
Record Dates: First submitted 2019-03-08; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Intervention Model Description: The clinical study is a randomized, double-blinded, controlled study aimed to assess the effect of zeolite-intervention in osteoporotic patients on the bone mineral density and bone turnover in comparison to osteoporotic patients control group that received the placebo over a period of for 12 months. The study population will consist of 100 patients with osteoporosis defined according BMD criteria: T score -2, 5 on the femoral neck, and, or T -2, 5 on L1-L5, who have not been treated before, or in whom privies treatment did not been successful, despite a gender or age. The Panaceo and Placebo groups will be divided into 50 and 50 patients.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zeolite (Active Comparator): 50 subjects receive the substance 3 times per day as powder
  Interventions: Device: zeolite
- cellulose (Placebo Comparator): 50 subjects receive the substance 3 times per day as powder
  Interventions: Device: cellulose

INTERVENTIONS:
Device: zeolite — given for a period of 12 months
  Arms: zeolite
Device: cellulose — given for a period of 12 months
  Arms: cellulose

SUMMARY:
This study investigates the effect of zeolite on bone mineral metabolism. The clinical parameters include bone mineral density, bone remodelling markers, fractures and fallings, the subjective evaluation of the overall health status and intensity of the musculoskeletal pain measured by VAS.

DETAILED DESCRIPTION:
Randomized, placebo-controlled, double-blind study. The Study lasts 12 months. Study Population: The study population will consist of 100 patients with osteoporosis defined according BMD (bone mineral density) criteria: T score -2, 5 on the femoral neck, and, or T -2, 5 on L1-L5, who has not been treated before, or in whom privies treatment did not been successful, despite a gender or age. Subjects will be randomized in each cohort to receive PMA-zeolite (Panaceo) or placebo (1:1). All of them will receive Vit D3 800 j daily.

The double blind design can be reached by a "third party blinding" where a qualified person, not being involved in the assessment of the study, will administer the study treatment.

Follow up DXA, Ca, P, ALP, Osteocalcin, Cross laps, Creatinin will be done to each subject before the treatment, 6 months later and after 12 months. IVA (vertebral deformity assessment) will be performed before the treatment and after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 100 subjects with osteoporosis Among those, as a subgroup, 20 subjects with diabetes type 2 and osteoporosis

  * The osteoporosis- was diagnosed by standard DXA measurement (BMD T-score: - 2.5 or below )

Exclusion Criteria:

* chronic renal failure, secondary osteoporosis

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Change of BMD (Bone mineral density) | 0-6-12 months
  BMD measurements are used to see how well osteoporosis treatments are working

SECONDARY OUTCOMES:
Cange of Bone remodelling marker Osteocalcin | 0-6-12 months
  Osteocalcin- parameter of the bone formation rate
Cange of Bone remodelling marker Betacross laps | 0-6-12 months
  Betacross laps - parameter of the bone degradation rate

OTHER OUTCOMES:
Fractures and fallings | 12 months
  Fracture: evaluation if yes) or no) Falling: Fracture as a consequence OR no fracture OR no fallings reported
Intensity of the musculoskeletal pain measured by VAS | 0-12 months
  the scale based on patient's subjective evaluation at the beginning and at the end of the study.
Subjective evaluation of the overall health status and 6. | 0-12 months
  upon the end of the study in comparison to the beginning

REFERENCES:
- [Derived] Kraljevic Pavelic S, Saftic Martinovic L, Simovic Medica J, Zuvic M, Perdija Z, Krpan D, Eisenwagen S, Orct T, Pavelic K. Clinical Evaluation of a Defined Zeolite-Clinoptilolite Supplementation Effect on the Selected Blood Parameters of Patients. Front Med (Lausanne). 2022 May 27;9:851782. doi: 10.3389/fmed.2022.851782. eCollection 2022. PMID 35712111
- [Derived] Kraljevic Pavelic S, Micek V, Bobinac D, Bazdulj E, Gianoncelli A, Krpan D, Zuvic M, Eisenwagen S, Stambrook PJ, Pavelic K. Treatment of osteoporosis with a modified zeolite shows beneficial effects in an osteoporotic rat model and a human clinical trial. Exp Biol Med (Maywood). 2021 Mar;246(5):529-537. doi: 10.1177/1535370220968752. Epub 2020 Nov 12. PMID 33183068